CLINICAL TRIAL: NCT06949137
Title: A Single-center, Open-label, Single-arm, 3+3 Dose-escalation Phase I Clinical Study to Evaluate Safety and Tolerability of HMM910(Human Mesenchymal Stem Cells Injection) in Postmenopausal Women With Osteoporosis and at High Risk of Fracture
Brief Title: Intravenous Infusion of Human Mesenchymal Stem Cells (HMM910 ) in Postmenopausal Women With Osteoporosis at High Risk of Fracture
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Help Therapeutics (Industry)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JL , HL
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-04

CONDITIONS: Osteoporosis in Post-menopausal Women; Osteoporosis
Keywords: mesenchymal stem cell; osteooprpsis; post menopausal; intravenous; fracture; HMM910
MeSH Terms: conditions — Osteoporosis; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Dose Group (Experimental): 6.0×10^7
  Interventions: Biological: Human Umbilical Cord-derived Mesenchymal stem cell
- Medium Dose Group (Experimental): 1.2×10^8
  Interventions: Biological: Human Umbilical Cord-derived Mesenchymal stem cell
- High Dose Group (Experimental): 2.4×10^8
  Interventions: Biological: Human Umbilical Cord-derived Mesenchymal stem cell

INTERVENTIONS:
Biological: Human Umbilical Cord-derived Mesenchymal stem cell — Intravenous infusion of human mesenchymal stem cells (HMM910 ) at 20-25 drops per minute
  Other Names: HMM910

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of human umbilical cord-derived mesenchymal stem cells for injection (HMM910 ) in postmenopausal women with osteoporosis who are at high risk of fracture.

ELIGIBILITY:
Inclusion Criteria:

All of the following criteria must be met for inclusion:

1. Willingness to participate in the clinical trial and signing of informed consent;
2. Female, age between 45 (inclusive) and 85 (inclusive) years, with primary menopause for ≥2 years;
3. Body weight ≥40 kg, and body mass index (BMI) between 18 kg/m² (inclusive) and 30 kg/m² (inclusive);
4. Those who meet the diagnostic criteria for osteoporosis and have one of the following conditions: ① Fragile fracture occurred in the past 2 years; ② Suffered a fracture while receiving anti-osteoporosis medication; ③ History of multiple-site fractures (including vertebral, hip, proximal humerus, or distal radius, etc.); ④ Bone mineral density (BMD) T-score < -3.0 at the lumbar spine (L1-L4) or hip (total hip or femoral neck) as measured by DXA; ⑤ High risk of falling; ⑥ Calculated by FRAX (Fracture Risk Assessment Tool), a 10-year risk of major osteoporotic fracture >30% or hip fracture risk >4.5%; ⑦ Currently using medications known to cause skeletal harm [such as high-dose glucocorticoids (prednisolone ≥7.5 mg/day for over 3 months), etc.].

Exclusion Criteria：

Subjects who meet one or more of the following criteria will be excluded:

1. Diseases affecting bone metabolism: various metabolic bone diseases such as osteogenesis imperfecta and osteomalacia; Paget's disease of bone, hypercalcemia, hypocalcemia (participants must not have used calcium supplements within 24 hours before blood sampling for serum calcium screening); Cushing's syndrome, hyperprolactinemia; hypopituitarism; acromegaly, etc.; hyperparathyroidism or hypoparathyroidism; secondary menopause, etc.
2. Secondary osteoporosis and other severe conditions, such as primary bone tumors (e.g., multiple myeloma, osteosarcoma, chondrosarcoma), secondary bone tumors, hematologic malignancies, or drug-induced osteoporosis.
3. Current malignancy, history of malignancy not cured for at least 5 years, or disability due to severe or long-term diseases (such as stroke, Parkinson's disease, multiple sclerosis) resulting in inability to ambulate.
4. Severe infectious diseases, autoimmune diseases (e.g., systemic lupus erythematosus), uncontrolled severe hypertension, or diabetes mellitus with severe complications or unstable blood glucose; severe cardiovascular, cerebrovascular, or other significant diseases.
5. Allergic constitution: known allergy to products derived from mammalian cells or to the investigational product of clinical significance.
6. Patients who have undergone major organ or bone marrow transplantation; patients who have received external radiation or skeletal implantation of radioactive materials.
7. Patients who have previously received any form of cell therapy.
8. Previous treatment with anti-osteoporosis drugs or medications affecting bone metabolism: ① Treatment with any PTH analog within the past 6 months (including participation in clinical trials of similar products); ② Treatment with any RANKL inhibitor (such as denosumab) within the past year; ③ Cumulative use of oral bisphosphonates for ≥3 years; or cumulative use >3 months but <3 years with the last dose administered within 6 months before screening, or intravenous bisphosphonate use within 24 months before screening.
9. DXA measurement: ① Fewer than two lumbar vertebrae were measurable by DXA; ② Height, weight, or body size may impede accurate DXA measurement.
10. HBV-DNA ≥1,000 copies (cps)/mL or above the upper limit of normal; hepatitis C virus (HCV) antibody positive and HCV RNA copies above the upper limit of normal; positive syphilis antibody, or HIV antibody.
11. Malabsorption syndromes, such as Crohn's disease and chronic pancreatitis. Known impaired absorption of calcium or vitamin D.
12. History of neurological or psychiatric disorders.
13. Current uncontrolled thyroid disease, hyperthyroidism, or hypothyroidism; thyroid stimulating hormone (TSH) level below normal range; TSH elevated (>5.5 μIU/mL but ≤10.0 μIU/mL) and serum T4 outside the normal range; TSH >10.0 μIU/mL.
14. Known severe hepatic insufficiency (AST or ALT ≥2×ULN, ALP or total bilirubin ≥1.5×ULN), liver cirrhosis, unstable liver disease, or known clinically significant biliary anomalies as judged by the investigator (excluding Gilbert's syndrome or asymptomatic gallstones); known moderate to severe chronic kidney disease (eGFR <60 mL/min/1.73 m²).
15. Evidence of alcohol abuse or drug abuse within 12 months before screening, as determined by the investigator, may interfere with the understanding or completion of the study by the participant.
16. Participation in another clinical trial within 6 months before screening.
17. Other conditions deemed by the investigator as unsuitable for participation.

Ages: 45 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-03-06 (Estimated); Study Completion 2026-09-06 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Treatment-Related Adverse Events | Within 4 weeks after administration
  Any adverse reactions/adverse events (AEs) related to MSC treatment occurring within 4 weeks after the completion of MSC administration in all subjects, and their severity (graded according to CTCAE criteria).

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Assessment of hMSC100 Target Gene Levels | From enrollment to the end of treatment at 20 weeks
  To evaluate the pharmacokinetic profile of hMSC100, the levels of the hMSC100 target gene will be measured at various time points before and after stem cell treatment. PK parameters will be calculated if data allows.
Change from Baseline in Bone Turnover Markers and Estrogen Levels | Bone turnover markers: At Day 3, and Weeks 1, 2, 4, 8, 16, and 20 after the first treatment. Estrogen levels: At Weeks 2, 4, and 20 after the first treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Li, MD, PhD, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School; Hua Lin, MD, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- HELP Therapeutics, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Results of the trial will be disseminated to study participants through direct consultation with a trial clinician at completion of the trial, as well as through the publication of results.
Supporting Information: Study Protocol, CSR
Time Frame: One year after study completed
Access Criteria: Results of the trial will be disseminated to study participants through direct consultation with a trial clinician at completion of the trial, as well as through the publication of results.